CLINICAL TRIAL: NCT04219709
Title: Brain Function, Cognition, and Hypoglycemia Tolerance in Patients With Type 1 Diabetes Mellitus in the Setting of Nutritional Ketosis Versus Standard Carbohydrate Diet
Brief Title: Effects of Ketosis on Brain Function in Patients With T1DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Belinda Lennerz, Instructor in Pediatric Endocrinology, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00030039_2
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Type1diabetes
Keywords: nutrition; very low carbohydrate diet; ketogenic diet; nutritional ketosis; cognitive function; brain; metabolism; ketones; ketosis
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a parallel design to receive a standard carbohydrate diet versus very low carbohydrate diet. Both of diet groups will undergo euglycemic-hypoglycemic insulin clamps and MRI studies to assess brain hypoglycemia tolerance. The standard diet group will undergo an additional euglycemic-hypoglycemic insulin clamp - with and without exogenous oral ketones in random order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very low carbohydrate diet (Experimental): Dietary Intervention, food delivery
  Interventions: Other: Very low carbohydrate diet
- Standard diet (Active Comparator): Dietary Intervention, food delivery
  Interventions: Other: Standard carbohydrate diet

INTERVENTIONS:
Other: Very low carbohydrate diet — All meals will be delivered and participants will consume study foods exclusively. Participants will receive a fiber supplement with each meal as needed to promote digestive health, and a daily multi-vitamin, magnesium and omega-3 supplement to ascertain micronutrient sufficiency. Participants will be weighed at each study visit and the diet plan will be adjusted for satiety and weight-maintenance.
  The diet composition will be as follows: 5% carbohydrate, 75% fat, 20% protein.
  Arms: Very low carbohydrate diet
Other: Standard carbohydrate diet — All meals will be delivered and participants will consume study foods exclusively. Participants will receive a daily multi-vitamin and omega-3 supplement to ascertain micronutrient sufficiency. Participants will be weighed at each study visit and the diet plan will be adjusted for satiety and weight-maintenance.
  The diet composition will be as follows: 50% carbohydrate, 30% fat, 20% protein.
  Arms: Standard diet

SUMMARY:
The scientific goal of this study is to examine the effects of a ketogenic diet on hypoglycemia tolerance and brain function in people with type 1 diabetes mellitus (T1D) and to clarify the mechanistic role of ketones in this process. Glycemic management of T1D is typified by alternating periods of hyper- and hypo-glycemia. Because brain metabolism under usual conditions depends on glucose, acute hypoglycemia leads to immediate complications including impaired cognitive function and a counter-regulatory hormone response. Recurrent hypoglycemia is associated with functional and structural changes in the brain and contributes to the cognitive decline observed in individuals with diabetes. The state of nutritional ketosis (as it occurs during fasting or when following a ketogenic [very low carbohydrate] diet) may protect against these acute and chronic complications. As the body relies on fat metabolism, ketone bodies build up and provide an alternative fuel for the brain. Studies during hypoglycemia have shown better cognitive function and less hypoglycemia symptoms in the setting of nutritional ketosis or with ketone administration. This physiological benefit may have special relevance for people with T1D who experience hypoglycemia frequently. To date, no mechanistic studies have examined brain effects of nutritional ketosis in T1D; nor have any trials explored the potential relevance of this for diabetes care.

DETAILED DESCRIPTION:
To test the hypothesis that a ketogenic diet increases hypoglycemia tolerance and improves brain function and cognitive performance during hypoglycemia, the researchers propose a randomized mechanistic study using insulin infusions and neuroimaging. The study will leverage an existing randomized controlled trial (RCT) in 32 young adults with T1D who will receive a ketogenic vs a standard carbohydrate diet for 12 weeks. Researchers will conduct a euglycemic-hypoglycemic insulin clamp using a continuous infusion of insulin, along with a glucose infusion that is adjusted to keep blood glucose levels normal (90 mg/dL), followed by a slow drop to hypoglycemia (50 mg/dL). Researchers will assess activation and connectivity of relevant brain areas by magnetic resonance imaging (MRI). Using continuous imaging during the gradual glycemic descent from 90 mg/dL to 50 mg/dL, the researchers will establish the glycemic threshold at which the hypothalamus becomes activated. Using a combination of MRI modalities, they will assess brain activation and connectivity changes during hypoglycemia versus euglycemia, both during rest and in relation to a cognitive task. Brain findings will be integrated with physiologic (blood levels of glucose, ketones, free fatty acids, counter-regulatory hormones) and behavioral (reaction time, cognitive task performance, hypoglycemia symptoms scale) parameters. In additional studies, researchers will give an oral ketone drink to raise blood ketone levels in participants in the standard carbohydrate diet arm. They will perform the same insulin infusion and MRI investigations to clarify the mechanistic role of ketones in mediating brain activation patterns. Comparison will be between nutritional vs no ketosis, exogenous vs no ketosis, and nutritional vs exogenous ketosis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with T1D for at least 1 year
* Age 18 to 40 years
* Tanner stage ≥ IV
* BMI 18.5-35 kg/m2
* Stable glycemic control (HbA1c 6.5-9%)
* Use of a continuous glucose monitor (CGM)
* Use of an insulin pump
* Attendance of at least 1 diabetes care visit over the past 12 months (including virtual)

Exclusion Criteria:

* Ketoacidosis or severe hypoglycemia with seizure or coma in the past 6 months
* Dietary restrictions or intolerances that are incompatible with the planned food deliveries, e.g. celiac disease, gastroparesis, certain food allergies
* Following a weight-loss or otherwise restrictive diet
* Vigorous exercise >2 hours on >3 days a week
* History of an eating disorder or at risk for eating disorder, assessed by the Eating Disorders Diagnostic Scale (EDDS)
* Major medical illness or use of medications other than insulin and metformin that could interfere with metabolic or glycemic variables
* Significant psychiatric illness
* Smoking, use of recreational drugs, or excessive alcohol consumption
* Pregnancy or breastfeeding
* Anemia
* For participants who undergo MRI:

  1. Standard MRI exclusion criteria
  2. Irregular menses
  3. Use of psychotropic medication other than SSRIs or other mild antidepressant or anxiety medications (unless these medications are safe to be held for several days to allow for the acquisition of MRI data).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic threshold for hypothalamic activation | Diet week 5-12
  The blood glucose level at which hypothalamic activation is detected by continuous BOLD functional MRI during a 40 min glycemic descent from 90 to 50 mg/dL

SECONDARY OUTCOMES:
Resting brain activation changes in brain areas related to cognition during hypoglycemia | Diet week 5-12
  Resting brain activation will be measured by arterial spin labeling (ASL) during euglycemia and hypoglycemia and differences will be reported
Task-related brain activation changes during hypoglycemia in brain areas related to cognition | Diet week 5-12
  Task-related brain activation will be measured during a working memory task (n-back) by BOLD during euglycemia and hypoglycemia and differences will be reported
Functional connectivity changes in brain areas related to cognition during hypoglycemia | Diet week 5-12
  Functional connectivity activation will be measured using resting state functional MRI during euglycemia and hypoglycemia and differences will be reported
Response time changes during hypoglycemia | Diet week 5-12
  Response time to a working-memory cognitive task (n-back) will be measured during hypoglycemia and compared to the response time in euglycemia
Cognitive performance during hypoglycemia | Diet week 5-12
  Response accuracy of a cognitive task (n-back) during hypoglycemia compared to euglycemia will be reported
Hypoglycemia symptoms | Diet week 5-12
  A Hypoglycemia Symptoms Scale comprising 6 autonomic/neurogenic (sweating, palpitations, trembling, weakness, nausea, and hunger) and 5 neuroglycopenic (drowsiness, confusion, difficulty concentrating, lightheadedness, and headache) symptoms will be used to assess each symptom on a 0-4 scale (higher scores indicate more symptoms) during euglycemia and hypoglycemia. Average scores for hypoglycemia symptoms overall, autonomic/neurogenic symptoms, and neuroglycopenic symptoms will be reported for each time point.
Blood glucose level at which participant reports symptoms of hypoglycemia. | Diet week 5-12
  Participants will be instructed to push a response button when they first notice any symptoms of hypoglycemia during the glycemic descent phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No